CLINICAL TRIAL: NCT00464815
Title: Primary Vaccination Study in Subjects Aged 11-17 Years to Demonstrate the Non-inferiority of GSK Biologicals' Meningococcal Vaccine GSK134612 Vaccine Versus Mencevax™ ACWY
Brief Title: Non-Inferiority of Meningococcal Vaccine GSK134612 Versus Mencevax™ in 11-17 Year-Old Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109069
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-03

CONDITIONS: Infections, Meningococcal
Keywords: immunogenicity; safety; meningococcal vaccine
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Group A (Experimental): Subjects of 11-17 years of age who will receive GSK134612
  Interventions: Biological: Meningococcal vaccine GSK134612
- Group B (Active Comparator): Subjects of 11-17 years of age who will receive MencevaxTM ACWY
  Interventions: Biological: Mencevax™ ACWY

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — One intramuscular dose
  Arms: Group A
Biological: Mencevax™ ACWY — One subcutaneous dose
  Arms: Group B

SUMMARY:
The purpose of this study is to demonstrate, in 11-17 year old subjects, the non-inferiority of meningococcal vaccine GSK134612 compared to licensed meningococcal vaccine Mencevax™.

DETAILED DESCRIPTION:
Multicentre study with 2 treatment groups. Each subject will have 2 blood samples taken for immunogenicity analyses, one prior to vaccination and one taken 30 days later.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 11 and 17 years of age at the time of the vaccination.
* Written informed assent/consent obtained from the subject/ from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of the subject's/the subject's parent's/guardian's knowledge.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for two months after vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the dose of vaccine.
* Previous vaccination with meningococcal polysaccharide vaccine of serogroup A, C, W-135 and/or Y within the last five years.
* Previous vaccination with meningococcal polysaccharide conjugate vaccine of serogroup A, C, W-135 and/or Y.
* Previous vaccination with tetanus toxoid within the last month.
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1025 (Actual)
Dates: Start 2007-05-02 (Actual); Primary Completion 2008-04-16 (Actual); Study Completion 2008-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- India (4):
  - GSK Investigational Site, Goa
  - GSK Investigational Site, Indore
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
- GSK Investigational Site, City of Muntinlupa, Philippines
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tao Yuan County

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bermal N, Huang LM, Dubey AP, Jain H, Bavdekar A, Lin TY, Bianco V, Baine Y, Miller JM. Safety and immunogenicity of a tetravalent meningococcal serogroups A, C, W-135 and Y conjugate vaccine in adolescents and adults. Hum Vaccin. 2011 Feb;7(2):239-47. doi: 10.4161/hv.7.2.14068. Epub 2011 Feb 1. PMID 21343698
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 109069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The target sample size was 1024 enrolled subjects, but a total of 1025 subjects (in all age strata) were actually enrolled and vaccinated in seven study centres in India, Taiwan and the Philippines.
Groups:
- Nimenrix Group: Healthy male and female subjects aged 11 through 17 years, who received 1 dose of Nimenrix (GSK134612) vaccine, administered intramuscularly into the deltoid region of the non-dominant arm.
- Mencevax ACWY Group: Healthy male and female subjects aged 11 through 17 years, who received 1 dose of Mencevax ACWY vaccine, administered subcutaneously into the non-dominant upper arm.
Period: Overall Study
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Started | 768 | 257
Completed | 762 | 254
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix Group | Mencevax ACWY Group | Total
Number analyzed (Participants) | 768 | 257 | 1025
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.3 (1.97) | 14.3 (1.97) | 14.3 (1.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 414 | 135 | 549
  Male | 354 | 122 | 476
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian-Central/South Asian heritage | 296 | 100 | 396
  Geographic ancestry: Asian-East Asian heritage | 175 | 59 | 234
  Geographic ancestry: Asian-South East Asian heritage | 297 | 98 | 395

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Response to Meningococcal Antigens
Description: Vaccine response induced by Neisseria meningitidis serogroups A, C, W-135 and Y (MenA, MenC, MenW-135 and menY) as measured by serum bactericidal antibodies using baby rabbit complement (rSBA), was defined as an rSBA titer of at least 1:32 in subjects initially seronegative [rSBA titer below (<) 1:8] and as a 4-fold increase in titer in subjects initially seropositive [rSBA titer greater than or equal to (≥) 1:8].
Time Frame: One month post-vaccination (At Month 1)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variable measures and assay results were available for antibodies against at least one study vaccine antigen component.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 657 | 219
Participants
  rSBA-MenA: number analyzed (Participants) | 553 | 191
  rSBA-MenA | 472 | 148
  rSBA-MenC: number analyzed (Participants) | 642 | 211
  rSBA-MenC | 625 | 204
  rSBA-MenW-135: number analyzed (Participants) | 639 | 216
  rSBA-MenW-135 | 616 | 189
  rSBA-MenY | 616 | 172
Statistical Analysis 1: Comparison: Nimenrix Group vs Mencevax ACWY Group; To demonstrate the non-inferiority of Nimenrix vaccine versus Mencevax ACWY vaccine in term of rSBA-MenA vaccine response, the standardized asymptotic 95% CI for the difference in rSBA vaccine response rate for the meningococcal serogroup A (Nimenrix Group rate minus Mencevax ACWY Group rate) one month after vaccination was computed; Test type: Non-Inferiority — Criterion for non-inferiority: the lower limit (LL) of the 2-sided standardized asymptotic 95% confidence interval (CI) for the group difference (Nimenrix Group minus Mencevax ACWY Group) in the percentage of subjects with bactericidal vaccine response was greater than or equal to (≥) the pre-defined clinical limit of -10%; Rate difference = 7.87, 95% CI 2-sided [1.63 to 14.87]
Statistical Analysis 2: Comparison: Nimenrix Group vs Mencevax ACWY Group; To demonstrate the non-inferiority of Nimenrix vaccine versus Mencevax ACWY vaccine in term of rSBA-MenC vaccine response, the standardized asymptotic 95% CI for the difference in rSBA vaccine response rate for the meningococcal serogroup C (Nimenrix Group rate minus Mencevax ACWY Group rate) one month after vaccination was computed; Test type: Non-Inferiority — Criterion for non-inferiority: the lower limit (LL) of the 2-sided standardized asymptotic 95% confidence interval for the group difference [Nimenrix Group minus Mencevax ACWY Group] in the percentage of subjects with bactericidal vaccine response was greater than or equal to (≥) the pre-defined clinical limit of -10%; Rate Difference = 0.67, 95% CI 2-sided [-1.65 to 4.18]
Statistical Analysis 3: Comparison: Nimenrix Group vs Mencevax ACWY Group; To demonstrate the non-inferiority of Nimenrix vaccine versus Mencevax ACWY vaccine in term of rSBA-MenW-135 vaccine response, the standardized asymptotic 95% CI for the difference in rSBA vaccine response rate for the meningococcal serogroup W-135 (Nimenrix Group rate minus Mencevax ACWY Group rate) one month after vaccination was computed; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Rate difference = 8.9, 95% CI 2-sided [4.78 to 14.14]
Statistical Analysis 4: Comparison: Nimenrix Group vs Mencevax ACWY Group; To demonstrate the non-inferiority of Nimenrix vaccine versus Mencevax ACWY vaccine in term of rSBA-MenY vaccine response, the standardized asymptotic 95% CI for the difference in rSBA vaccine response rate for the meningococcal serogroup Y (Nimenrix Group rate minus Mencevax ACWY Group rate) one month after vaccination was computed; Test type: Non-Inferiority — Criterion for non-inferiority: the lower limit (LL) of the 2-sided standardized asymptotic 95% confidence interval (CI) for the group difference [Nimenrix Group minus Mencevax ACWY Group] in the percentage of subjects with bactericidal vaccine response was greater than or equal to (≥) the pre-defined clinical limit of -10%; Rate difference = 15.22, 95% CI 2-sided [9.89 to 21.37]

2. Primary Outcome: Number of Subjects With Any Grade 3 General (Solicited and Unsolicited) Symptoms
Description: General symptoms assessed included fatigue, fever (defined as axillary temperature), gastrointestinal symptoms and headache. Grade 3 symptom= event that prevented normal activities. Grade 3 fever= temperature above (>) 39.5 degrees Celsius (°C).
Time Frame: During the 4-day (Days 0-3) period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 768 | 257
Participants | 12 | 1
Statistical Analysis 1: Comparison: Nimenrix Group vs Mencevax ACWY Group; To demonstrate the non-inferiority of Nimenrix™ vaccine versus Mencevax™ vaccine in terms of incidence of any Grade 3 general (solicited and unsolicited) symptom, the 2-sided standardised asymptotic 95% CI for the ratio between Nimenrix and Mencevax groups (Nimenrix over Mencevax) in the percentage of subjects with any grade 3 general symptom within 4 days after vaccination was computed for the safety analysis in study MenACWY-TT-036; Test type: Non-Inferiority — Criterion for non-inferiority: the upper limit (UL) of the 2-sided standardized asymptotic 95% CI for the ratio of the percentages of subjects with any Grade 3 general symptom was lower than or equal to (≤) the pre-defined clinical limit of 3.0; p = 0.1456, Chi-squared; Risk Ratio (RR) = 4.02, 95% CI 2-sided [0.68 to 24.6]

3. Secondary Outcome: Number of Subjects With rSBA-Men Antibody Titers ≥ the Cut-off Values
Description: Neisseria meningitidis serogroups A, C, W-135 and Y were measured by serum bactericidal assay using baby rabbit complement (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY). The cut-off values for the rSBA titers was greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: Prior to (Month 0) and one month after vaccination (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 678 | 224
Participants
  rSBA-MenA, Month 0 ≥ 1:8: number analyzed (Participants) | 557 | 191
  rSBA-MenA, Month 0 ≥ 1:8 | 463 | 148
  rSBA-MenA, Month 0 ≥ 1:128: number analyzed (Participants) | 557 | 191
  rSBA-MenA, Month 0 ≥ 1:128 | 427 | 128
  rSBA-MenA, Month 1 ≥ 1:8: number analyzed (Participants) | 674 | 224
  rSBA-MenA, Month 1 ≥ 1:8 | 674 | 223
  rSBA-MenA, Month 1 ≥ 1:128: number analyzed (Participants) | 674 | 224
  rSBA-MenA, Month 1 ≥ 1:128 | 674 | 223
  rSBA-MenC, Month 0 ≥ 1:8: number analyzed (Participants) | 648 | 211
  rSBA-MenC, Month 0 ≥ 1:8 | 381 | 121
  rSBA-MenC, Month 0 ≥ 1:128: number analyzed (Participants) | 648 | 211
  rSBA-MenC, Month 0 ≥ 1:128 | 277 | 79
  rSBA-MenC, Month 1 ≥ 1:8: number analyzed (Participants) | 673 | 224
  rSBA-MenC, Month 1 ≥ 1:8 | 673 | 224
  rSBA-MenC, Month 1 ≥ 1:128: number analyzed (Participants) | 673 | 224
  rSBA-MenC, Month 1 ≥ 1:128 | 672 | 223
  rSBA- MenW-135, Month 0 ≥ 1:8: number analyzed (Participants) | 640 | 216
  rSBA- MenW-135, Month 0 ≥ 1:8 | 519 | 176
  rSBA- MenW-135, Month 0 ≥ 1:128: number analyzed (Participants) | 640 | 216
  rSBA- MenW-135, Month 0 ≥ 1:128 | 373 | 120
  rSBA- MenW-135, Month 1 ≥ 1:8 | 677 | 224
  rSBA- MenW-135, Month 1 ≥ 1:128 | 677 | 223
  rSBA-MenY, Month 0 ≥ 1:8: number analyzed (Participants) | 659 | 219
  rSBA-MenY, Month 0 ≥ 1:8 | 597 | 186
  rSBA-MenY, Month 0 ≥ 1:128: number analyzed (Participants) | 659 | 219
  rSBA-MenY, Month 0 ≥ 1:128 | 538 | 167
  rSBA-MenY, Month 1 ≥ 1:8: number analyzed (Participants) | 677 | 224
  rSBA-MenY, Month 1 ≥ 1:8 | 677 | 224
  rSBA-MenY, Month 1 ≥ 1:128: number analyzed (Participants) | 677 | 224
  rSBA-MenY, Month 1 ≥ 1:128 | 677 | 224

4. Secondary Outcome: Meningococcal rSBA Antibody Titers
Description: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY antibody titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to (Month 0) and one month after vaccination (Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 678 | 224
Titer
  rSBA-MenA, Month 0: number analyzed (Participants) | 557 | 191
  rSBA-MenA, Month 0 | 208.1 [176.4 to 245.5] | 155.9 [113.8 to 213.7]
  rSBA-MenA, Month 1: number analyzed (Participants) | 674 | 224
  rSBA-MenA, Month 1 | 5928.5 [5557.4 to 6324.3] | 2947.2 [2611.7 to 3325.7]
  rSBA-MenC, Month 0: number analyzed (Participants) | 648 | 211
  rSBA-MenC, Month 0 | 44.1 [37.3 to 52.2] | 40.9 [30.2 to 55.3]
  rSBA-MenC, Month 1: number analyzed (Participants) | 673 | 224
  rSBA-MenC, Month 1 | 13109.8 [11939.1 to 14395.2] | 8222 [6807.5 to 9930.4]
  rSBA- MenW-135, Month 0: number analyzed (Participants) | 640 | 216
  rSBA- MenW-135, Month 0 | 109.4 [94.6 to 126.6] | 112.2 [87.2 to 144.3]
  rSBA- MenW-135, Month 1 | 8246.6 [7638.8 to 8902.7] | 2632.7 [2299.3 to 3014.4]
  rSBA-MenY, Month 0: number analyzed (Participants) | 659 | 219
  rSBA-MenY, Month 0 | 348.3 [303.5 to 399.7] | 299 [225.2 to 397]
  rSBA-MenY, Month 1: number analyzed (Participants) | 677 | 224
  rSBA-MenY, Month 1 | 14086.5 [13168 to 15069] | 5066.3 [4463.1 to 5750.9]

5. Secondary Outcome: Number of Subjects With Anti-tetanus Toxoid (Anti-TT) Greater Than (>) the Cut-off Value
Description: The cut-off value of the assay was an anti-tetanus toxoid antibody titer greater than (>) 0.1 international units per milliliter (IU/mL).
Time Frame: Prior to (Month 0) and one month after vaccination (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 679 | 224
Participants
  Anti-TT, Month 0 | 439 | 155
  Anti-TT, Month 1 | 662 | 157

6. Secondary Outcome: Anti-TT Antibody Concentrations
Description: Antibody concentrations are presented as geometric mean concentrations (GMCs) and expressed in international units per milliliter (IU/mL).
Time Frame: Prior to (Month 0) and one month after vaccination (Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 679 | 224
IU/mL
  Anti-TT, Month 0 | 0.367 [0.321 to 0.419] | 0.41 [0.326 to 0.516]
  Anti-TT, Month 1 | 10.305 [9.131 to 11.631] | 0.459 [0.364 to 0.58]

7. Secondary Outcome: Number of Subjects With Anti-meningococcal Polysaccharides (PS) Antibody Concentrations ≥ the Cut-off Values
Description: The cut-off values of the assay was an anti-PS concentration greater than or equal to (≥) 0.3 micrograms per milliliter (μg/mL) and ≥ 2.0 μg/mL.
Time Frame: Prior to (Month 0) and one month after vaccination (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 347 | 114
Participants
  Anti-PSA ≥ 0.3 ug/mL, Month 0: number analyzed (Participants) | 322 | 102
  Anti-PSA ≥ 0.3 ug/mL, Month 0 | 235 | 75
  Anti-PSA ≥ 0.3 ug/mL, Month 1: number analyzed (Participants) | 341 | 107
  Anti-PSA ≥ 0.3 ug/mL, Month 1 | 341 | 107
  Anti-PSC ≥ 0.3 ug/mL, Month 0: number analyzed (Participants) | 335 | 108
  Anti-PSC ≥ 0.3 ug/mL, Month 0 | 50 | 21
  Anti-PSC ≥ 0.3 ug/mL, Month 1: number analyzed (Participants) | 331 | 107
  Anti-PSC ≥ 0.3 ug/mL, Month 1 | 331 | 107
  Anti-PSW-135 ≥ 0.3 ug/mL, Month 0: number analyzed (Participants) | 340 | 111
  Anti-PSW-135 ≥ 0.3 ug/mL, Month 0 | 40 | 8
  Anti-PSW-135 ≥ 0.3 ug/mL, Month 1: number analyzed (Participants) | 344 | 114
  Anti-PSW-135 ≥ 0.3 ug/mL, Month 1 | 340 | 113
  Anti-PSY ≥ 0.3 ug/mL, Month 0 | 49 | 16
  Anti-PSY ≥ 0.3 ug/mL, Month 1: number analyzed (Participants) | 342 | 114
  Anti-PSY ≥ 0.3 ug/mL, Month 1 | 342 | 113
  Anti-PSA ≥ 2 ug/mL, Month 0: number analyzed (Participants) | 322 | 102
  Anti-PSA ≥ 2 ug/mL, Month 0 | 130 | 40
  Anti-PSA ≥ 2 ug/mL, Month 1: number analyzed (Participants) | 341 | 107
  Anti-PSA ≥ 2 ug/mL, Month 1 | 341 | 107
  Anti-PSC ≥ 2 ug/mL, Month 0: number analyzed (Participants) | 335 | 108
  Anti-PSC ≥ 2 ug/mL, Month 0 | 17 | 10
  Anti-PSC ≥ 2 ug/mL, Month 1: number analyzed (Participants) | 331 | 107
  Anti-PSC ≥ 2 ug/mL, Month 1 | 324 | 106
  Anti-PSW-135 ≥ 2 ug/mL, Month 0: number analyzed (Participants) | 340 | 111
  Anti-PSW-135 ≥ 2 ug/mL, Month 0 | 9 | 3
  Anti-PSW-135 ≥ 2 ug/mL, Month 1: number analyzed (Participants) | 344 | 114
  Anti-PSW-135 ≥ 2 ug/mL, Month 1 | 327 | 106
  Anti-PSY ≥ 2 ug/mL, Month 0 | 12 | 8
  Anti-PSY ≥ 2 ug/mL, Month 1: number analyzed (Participants) | 342 | 114
  Anti-PSY ≥ 2 ug/mL, Month 1 | 336 | 111

8. Secondary Outcome: Anti-meningococcal Polysaccharide Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL).
Time Frame: Prior to (Month 0) and one month after vaccination (Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 347 | 114
μg/mL
  Anti-PSA, Month 0: number analyzed (Participants) | 322 | 102
  Anti-PSA, Month 0 | 1.05 [0.88 to 1.24] | 1.04 [0.77 to 1.39]
  Anti-PSA, Month 1: number analyzed (Participants) | 341 | 107
  Anti-PSA, Month 1 | 86.06 [75.35 to 98.29] | 44.06 [34.4 to 56.42]
  Anti-PSC, Month 0: number analyzed (Participants) | 335 | 108
  Anti-PSC, Month 0 | 0.21 [0.19 to 0.24] | 0.25 [0.2 to 0.3]
  Anti-PSC, Month 1: number analyzed (Participants) | 331 | 107
  Anti-PSC, Month 1 | 22.83 [20.42 to 25.52] | 43.24 [35.8 to 52.23]
  Anti-PSW-135, Month 0: number analyzed (Participants) | 340 | 111
  Anti-PSW-135, Month 0 | 0.18 [0.17 to 0.2] | 0.18 [0.16 to 0.21]
  Anti-PSW-135, Month 1: number analyzed (Participants) | 344 | 114
  Anti-PSW-135, Month 1 | 17.82 [15.34 to 20.7] | 13.22 [10.47 to 16.68]
  Anti-PSY, Month 0 | 0.2 [0.18 to 0.22] | 0.22 [0.18 to 0.28]
  Anti-PSY, Month 1: number analyzed (Participants) | 342 | 114
  Anti-PSY, Month 1 | 23.77 [20.95 to 26.98] | 17.97 [14.3 to 22.59]

9. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed included pain, redness and swelling. Any= incidence of a particular symptom regardless of intensity. Grade 3 symptoms= symptoms that prevented normal activity. Grade 3 swelling= swelling spreading beyond 50 millimeters (mm).
Time Frame: During the 4-day (Days 0-3) period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects who had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 763 | 254
Participants
  Any Pain | 200 | 68
  Grade 3 Pain | 6 | 0
  Any Redness | 94 | 16
  Grade 3 Redness | 2 | 0
  Any Swelling | 71 | 16
  Grade 3 Swelling | 9 | 0

10. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed included fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any= incidence of a particular symptom regardless of intensity or relationship to vaccination. Grade 3= event that prevented normal activities. Grade 3 fever= fever > 39.5 °C. Related= general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 4-day (Days 0-3) period after vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 763 | 254
Participants
  Any Fatigue | 109 | 36
  Grade 3 Fatigue | 7 | 1
  Related Fatigue | 83 | 26
  Any Fever (Axillary) | 55 | 13
  Grade 3 Fever | 3 | 0
  Related Fever | 42 | 10
  Any Gastrointestinal symptoms | 35 | 11
  Grade 3 Gastrointestinal symptoms | 0 | 1
  Related Gastrointestinal symptoms | 24 | 9
  Any Headache | 102 | 27
  Grade 3 Headache | 5 | 1
  Related Headache | 81 | 19

11. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 768 | 257
Participants | 72 | 26

12. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to study end (Month 6)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 768 | 257
Participants | 3 | 2

13. Secondary Outcome: Number of Subjects With Specific Adverse Events
Description: These events consist of specific categories of adverse events (AEs) which included rash (e.g. hives, idiopathic thrombocytopenia purpura, petechiae), new onset of chronic illness(es) (NOCIs) (e.g. autoimmune disorders, asthma, type I diabetes and allergies), conditions prompting emergency room (ER) visits or non-routine physician office visits (i.e. office visits not related to well-being care, vaccination, injury or common acute illnesses such as upper respiratory tract infections, otitis media, pharyngitis, gastroenteritis), any events related to lack of meningococcal vaccine efficacy (i.e. meningococcal disease).
Time Frame: Up to study end (Month 6)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax ACWY Group
Number analyzed (Participants) | 768 | 257
Participants
  Any Rash | 6 | 1
  Any NOCIs | 0 | 0
  Any ER visits | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general adverse events (AEs): during the 4-day (Days 0-3) period after vaccination. Unsolicited AEs: up to one month after vaccination (Month 1). SAEs and specific AEs: up to study end (Month 6).
Groups:
- Nimenrix Group: Healthy male and female subjects aged 11 through 17 years, who received 1 dose of Nimenrix™ (GSK134612) vaccine, administered intramuscularly into the deltoid region of the non-dominant arm.
- Mencevax ACWY Group: Healthy male and female subjects aged 11 through 17 years, who received 1 dose of Mencevax™ ACWY vaccine, administered subcutaneously into the non-dominant upper arm.
Arm/Group | Nimenrix Group | Mencevax ACWY Group
All-Cause Mortality (participants affected / at risk) | 0/768 | 0/257
Serious Adverse Events (participants affected / at risk) | 3/768 | 2/257
Other Adverse Events (participants affected / at risk) | 311/768 | 99/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix Group (N=768) | Mencevax ACWY Group (N=257)
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 0
Amoebic dysentery (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Peritoneal abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix Group (N=768) | Mencevax ACWY Group (N=257)
Pain (General disorders) | 200 | 68
Redness (General disorders) | 94 | 16
Swelling (General disorders) | 71 | 16
Fatigue (General disorders) | 109 | 36
Fever (General disorders) | 55 | 13
Headache (General disorders) | 102 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.